CLINICAL TRIAL: NCT00385255
Title: A Study to Evaluate Immunogenicity and Safety of Boostrix When Co-administered With Fluarix in Subjects 19 Years of Age and Older
Brief Title: Immunogenicity, Safety of GSKs Tdap Vaccine Boostrix When Coadministered With GSKs Influenza Vaccine Fluarix in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106323
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Acellular Pertussis; Diphtheria; Tetanus
Keywords: Immunogenicity,; Influenza; Co-administration,; Tdap,
MeSH Terms: conditions — Diphtheria; Tetanus; Influenza, Human | interventions — fluarix; Boostrix

ARMS (2):
- BOOSTRIX+FLUARIX GROUP (Experimental): Healthy male or female adults, aged between 19 to 64 years of age inclusive and 65 years or older, who received Boostrix® vaccine co-administered with Fluarix® vaccine at Day 0, injected intramuscularly in the left and right upper deltoid regions, respectively.
  Interventions: Biological: Fluarix®; Biological: Boostrix®
- FLUARIX BOOSTRIX GROUP (Experimental): Healthy male or female adults, aged between 19 to 64 years of age inclusive and 65 years or older, who received Fluarix® vaccine at Day 0 and Boostrix® vaccine at Month 1, both injected intramuscularly in the upper left deltoid region.
  Interventions: Biological: Fluarix®; Biological: Boostrix®

INTERVENTIONS:
Biological: Fluarix® — GSK Biologicals' inactivated influenza split virus vaccine.
Biological: Boostrix® — GSK Biologicals' tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine adsorbed, containing 0.3 mg aluminum.

SUMMARY:
The current study will provide information for the use of Boostrix concomitantly with influenza vaccine in adults aged 19-64 years. This study will also provide safety and immunogenicity data in a cohort of adults aged greater than or equal to 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults aged between 19 to 64 years, inclusive for the primary cohort), or aged 65 years or older (for the exploratory cohort), at the time of vaccination.

Exclusion Criteria:

* Administration of an influenza vaccine within six months prior to study entry
* Administration of a diphtheria-tetanus (Td) booster within the previous 5 years.
* Administration of a Tdap vaccine at any time prior to study entry.
* Administration of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding vaccination, or planned use during the entire study period.
* History of diphtheria and/or tetanus and/or pertussis disease.
* History of serious allergic reaction (e.g. anaphylaxis) following any other tetanus toxoid, diphtheria toxoid or pertussis-containing vaccine or influenza vaccine or any component of the study vaccines.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1726 (Actual)
Dates: Start 2006-10-23 (Actual); Primary Completion 2007-02-28 (Actual); Study Completion 2007-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (11):
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Weston WM, Chandrashekar V, Friedland LR, Howe B. Safety and immunogenicity of a tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis vaccine when co-administered with influenza vaccine in adults. Hum Vaccin. 2009 Dec;5(12):858-66. doi: 10.4161/hv.9961. Epub 2009 Dec 31. PMID 19838080
- [Background] Weston WM, Friedland LR, Wu X, Howe B. Vaccination of adults 65 years of age and older with tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine (Boostrix((R))): results of two randomized trials. Vaccine. 2012 Feb 21;30(9):1721-8. doi: 10.1016/j.vaccine.2011.12.055. Epub 2011 Dec 31. PMID 22212127
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 106323 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106323 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106323 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106323 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106323 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106323 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 1726 subjects originally enrolled in this study, 8 subjects (7 subjects from the 19-64 years of age cohort and 1 subject from the 65 years of age cohort) did not receive the study vaccine and hence were not included in the Total Vaccinated Cohort.
Period: Overall Study
Arm/Group | Boostrix+Fluarix Group | Fluarix Boostrix Group
Started | 860 | 858
≥ 65 Years of Age (YOA) Cohort | 112 | 109
19-64 Years of Age (YOA) Cohort | 748 | 749
Completed | 839 | 785
Not Completed | 21 | 73
Not completed — Serious Adverse Event | 1 | 2
Not completed — Protocol Violation | 0 | 4
Not completed — Withdrawal by Subject | 0 | 8
Not completed — Migrated/moved from study area | 0 | 1
Not completed — Lost to Follow-up | 20 | 58

BASELINE CHARACTERISTICS:
Groups:
- Boostrix+Fluarix Group: Healthy male or female adults, aged between 19 to 64 years inclusive and 65 years or older, who received Boostrix® vaccine co-administered with Fluarix® vaccine at Day 0, injected intramuscularly in the left and right upper deltoid regions, respectively.
- Fluarix Boostrix Group: Healthy male or female adults, aged between 19 to 64 years inclusive and 65 years or older, who received Fluarix® vaccine at Day 0 and Boostrix® vaccine at Month 1, both injected intramuscularly in the upper left deltoid region.
- Total: Total of all reporting groups
Arm/Group | Boostrix+Fluarix Group | Fluarix Boostrix Group | Total
Number analyzed (Participants) | 860 | 858 | 1718
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.95 (14.74) | 49.29 (14.58) | 49.12 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 527 | 481 | 1008
  Male | 333 | 377 | 710
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African heritage/African American | 69 | 82 | 151
  Geographic ancestry: American Indian or Alaskan native | 2 | 0 | 2
  Geographic ancestry: Asian-Central/South Asian heritage | 0 | 1 | 1
  Geographic ancestry: Asian-East Asian heritage | 1 | 2 | 3
  Geographic ancestry: Asian-Japanese heritage | 1 | 2 | 3
  Geographic ancestry: Asian-South East Asian heritage | 3 | 4 | 7
  Geographic ancestry: Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Geographic ancestry: White-Arabic/North African heritage | 7 | 4 | 11
  Geographic ancestry: White-Caucasian/European heritage | 759 | 747 | 1506
  Geographic ancestry: Not specified | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphteria (D) and Tetanus (T) Toxoid Antigens
Description: A seroprotected subject was defined as a vaccinated subject with anti-D and anti-T antibody concentrations equal to or above (≥) 0.1 International Units per milliliter (IU/mL), respectively.
Time Frame: At Month 1 post-Boostrix® vaccination
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Groups:
- Boostrix+Fluarix 19-64 YOA Group: Healthy male or female adults, between 19 to 64 years of age (YOA) inclusive, who received Boostrix® vaccine co-administered with Fluarix® vaccine at Day 0, injected intramuscularly in the left and right upper deltoid regions, respectively.
- Fluarix Boostrix 19-64 YOA Group: Healthy male or female adults, between 19 to 64 years of age (YOA) inclusive, who received Fluarix® vaccine at Day 0 and Boostrix® vaccine at Month 1, both injected intramuscularly in the upper left deltoid region.
- Boostrix+Fluarix ≥ 65 YOA Group: Healthy male or female adults, aged 65 years or older, who received Boostrix® vaccine co-administered with Fluarix® vaccine at Day 0, injected intramuscularly in the left and right upper deltoid regions, respectively.
- Fluarix Boostrix ≥ 65 YOA Group: Healthy male or female adults, aged 65 years or older, who received Fluarix® vaccine at Day 0 and Boostrix® vaccine at Month 1, both injected intramuscularly in the upper left deltoid region.
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 713 | 654 | 108 | 102
Participants
  Anti-D: number analyzed (Participants) | 712 | 653 | 106 | 98
  Anti-D | 677 | 614 | 93 | 79
  Anti-T | 700 | 653 | 105 | 95
Statistical Analysis 1: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in seroprotection rates against diphteria toxoid: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Boostrix® vaccine administered alone at Month 1 (Fluarix Boostrix 19-64 YOA Group), in terms of seroprotection rates for anti-D antibody, one month post-Boostrix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% confidence interval (CI) for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentages of subjects with anti-D antibody concentrations ≥ 0.1 IU/mL, being ≥ - 10%; Difference in percentage = 1.06, 95% CI 2-sided [-1.36 to 3.56]
Statistical Analysis 2: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in seroprotection rates against tetanus toxoid: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Boostrix® vaccine administered alone at Month 1 (Fluarix Boostrix 19-64 YOA Group), in terms of seroprotection rates for anti-T antibody, one month post-Boostrix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+ Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-T antibody concentrations ≥ 0.1 IU/mL, being ≥ - 10%; Difference in percentage = -1.67, 95% CI 2-sided [-2.96 to -0.74]

2. Primary Outcome: Number of Subjects With Anti-T Antibody Concentrations ≥ the Assay Cut-off Value
Description: The assay cut-off value was ≥ 1.0 IU/mL, as assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: At Month 1 post-Boostrix® vaccination
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity measures were available.
Measure: Count of Participants; unit: Participants
Groups:
- Boostrix+Fluarix 19-64 YOA Group: Healthy male or female adults, aged between 19 to 64 years inclusive, who received Boostrix® vaccine co-administered with Fluarix® vaccine at Day 0, injected intramuscularly in the left and right upper deltoid regions, respectively.
- Fluarix Boostrix 19-64 YOA Group: Healthy male or female adults, aged between 19 to 64 years inclusive, who received Fluarix® vaccine at Day 0 and Boostrix® vaccine at Month 1, both injected intramuscularly in the upper left deltoid region.
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 713 | 654 | 108 | 102
Participants | 687 | 621 | 94 | 84
Statistical Analysis 1: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in seropositivity rates against tetanus toxoid: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Boostrix® vaccine administered alone at Month 1 (Fluarix Boostrix 19-64 YOA Group), in terms of seropositivity rates for anti-T antibody, one month post-Boostrix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-T antibody concentrations ≥ 1.0 IU/mL, being ≥ - 10%; Difference in percentage = 1.40, 95% CI 2-sided [-0.77 to 3.68]

3. Primary Outcome: Antibody Concentrations Against Pertussis Toxoid (PT), Filamentous Hemagglutinin (FHA) and Pertactin (PRN) Antigens
Description: Anti-PT, anti-FHA and anti-PRN antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per milliliter (EL.U/mL).
Time Frame: At Month 1 post-Boostrix® vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 713 | 655 | 108 | 101
EL.U/mL
  Anti-PT: number analyzed (Participants) | 683 | 629 | 103 | 97
  Anti-PT | 57.5 [53.1 to 62.3] | 76.9 [71.1 to 83.2] | 51.2 [40.8 to 64.2] | 59.3 [47.0 to 74.8]
  Anti-FHA: number analyzed (Participants) | 712 | 654 | 107 | 100
  Anti-FHA | 467.6 [434.9 to 502.8] | 663.3 [613.3 to 717.4] | 502.5 [409.5 to 616.7] | 669.6 [539.1 to 831.8]
  Anti-PRN | 234.9 [208.7 to 264.3] | 343.6 [302.5 to 390.1] | 87.9 [60.1 to 128.5] | 97.0 [68.1 to 138.4]
Statistical Analysis 1: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in adjusted GMC ratios for anti-PT antibody: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Boostrix® vaccine administered alone at Month 1 (Fluarix Boostrix 19-64 YOA Group), in terms of geometric mean concentrations (GMCs) for anti-PT antibody, one month post-Boostrix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for GMC ratios of antibodies against the pertussis toxoid (PT) antigens between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group) being ≥ 0.67; ANCOVA; Adjusted GMC ratio = 0.74, 95% CI 2-sided [0.67 to 0.82]
Statistical Analysis 2: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in adjusted GMC ratio for anti-FHA antibody: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Boostrix® vaccine administered alone at Month 1 (Fluarix Boostrix 19-64 YOA Group), in terms of geometric mean concentrations (GMCs) for anti-FHA antibody, one month post-Boostrix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for GMC ratios of antibodies against the filamentous hemagglutinin (FHA) antigens between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group) being ≥ 0.67; ANCOVA; Adjusted GMC ratio = 0.71, 95% CI 2-sided [0.64 to 0.79]
Statistical Analysis 3: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in adjusted GMC ratio for anti-PRN antibody: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Boostrix® vaccine administered alone at Month 1 (Fluarix Boostrix 19-64 YOA Group), in terms of geometric mean concentrations (GMCs) for anti-PRN antibody, one month post-Boostrix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for GMC ratios of antibodies against the pertactin (PRN) antigens between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group) being ≥ 0.67; ANCOVA; Adjusted GMC ratio = 0.70, 95% CI 2-sided [0.60 to 0.81]

4. Primary Outcome: Number of Subjects With Serum Haemagglutinin Inhibition (HI) Titers Against 3 Strains of Influenza
Description: The antibody titer cut-off value for the 3 influenza strains assessed (H1N1, H3N2 and B) was ≥ 1:40.
Time Frame: At Month 1 post-Fluarix® vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 711 | 675 | 108 | 103
Participants
  Anti-H1N1 | 669 | 643 | 92 | 88
  Anti-H3N2 | 694 | 663 | 104 | 95
  Anti-B | 685 | 654 | 107 | 101
Statistical Analysis 1: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in percentage of subjects with anti-H1N1 antibody titers ≥ 1:40: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Fluarix® vaccine administered alone at Day 0 (Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-H1N1 antibody titers ≥ 1:40, one month post-Fluarix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-H1N1 antibody titers ≥ 1:40 being ≥ -10%; Difference in percentage = -1.17, 95% CI 2-sided [-3.58 to 1.23]
Statistical Analysis 2: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in percentage of subjects with anti-H3N2 antibody titers ≥ 1:40: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Fluarix® vaccine administered alone at Day 0 (Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-H3N2 antibody titers ≥ 1:40, one month post-Fluarix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-H3N2 antibody titers ≥ 1:40 being ≥ -10%; Difference in percentage = -0.61, 95% CI 2-sided [-2.22 to 0.96]
Statistical Analysis 3: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in percentage of subjects with anti-B antibody titers ≥ 1:40: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Fluarix® vaccine administered alone at Day 0 (Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-B antibody titers ≥ 1:40, one month post-Fluarix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with anti-B antibody titers ≥ 1:40 being ≥ -10%; Difference in percentage = -0.55, 95% CI 2-sided [-2.52 to 1.42]

5. Primary Outcome: Number of Seroconverted Subjects Against Influenza Antigens H1N1, H3N2, and B
Description: Seroconversion for HI antibodies is defined as: For initially seronegative subjects: post-vaccination antibody titer ≥ 1:40 at Month 1 post-Boostrix® vaccination; For initially seropositive subjects: antibody titer at Month 1≥ 4 fold the pre-vaccination antibody titer.
Time Frame: At Month 1 post-Fluarix® vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 708 | 672 | 108 | 102
Participants
  Anti-H1N1 | 414 | 377 | 37 | 32
  Anti-H3N2 | 560 | 494 | 72 | 64
  Anti-B | 463 | 425 | 41 | 43
Statistical Analysis 1: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in seroconversion rates for anti-H1N1 antibody: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Fluarix® vaccine administered alone at Day 0 (Fluarix Boostrix 19-64 YOA Group), in terms of seroconversion rates for anti-H1N1 antibody, one month post-Fluarix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with ≥ 4-fold increase in anti-H1N1 antibody titers (seroconversion) being ≥ -10%; Difference in seroconversion rate = 2.37, 95% CI 2-sided [-2.84 to 7.58]
Statistical Analysis 2: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in seroconversion rates for anti-H3N2 antibody: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Fluarix® vaccine administered alone at Day 0 (Fluarix Boostrix 19-64 YOA Group), in terms of seroconversion rates for anti-H3N2 antibody, one month post-Fluarix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with ≥ 4-fold increase in anti-H3N2 antibody titers (seroconversion) being ≥ -10%; Difference in seroconversion rate = 5.58, 95% CI 2-sided [1.10 to 10.07]
Statistical Analysis 3: Comparison: Boostrix+Fluarix 19-64 YOA Group vs Fluarix Boostrix 19-64 YOA Group; Difference in seroconversion rates for anti-B antibody: To demonstrate that the immunogenicity of Boostrix® vaccine co-administered with Fluarix® vaccine (Boostrix+Fluarix 19-64 YOA Group) at Day 0, was non-inferior to that of Fluarix® vaccine administered alone at Day 0 (Fluarix Boostrix 19-64 YOA Group), in terms of seroconversion rates for anti-B antibody, one month post-Fluarix® vaccination; Test type: Non-Inferiority — Non-inferiority was defined as the lower limit of the 95% CI for the difference between the two groups (Boostrix+Fluarix 19-64 YOA Group minus Fluarix Boostrix 19-64 YOA Group), in terms of percentage of subjects with ≥ 4-fold increase anti-B antibody titers (seroconversion) being ≥ -10%; Difference in seroconversion rate = 2.15, 95% CI 2-sided [-2.90 to 7.20]

6. Secondary Outcome: Number of Seropositive Subjects With Anti-D Antibody Concentrations Above the Cut-off Value
Description: A seropositive subject was a subject whose antibody concentration was greater than or equal (≥) to the cut-off value of 1.0 IU/mL.
Time Frame: At Month 1 post-Boostrix® vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 712 | 653 | 106 | 98
Participants | 579 | 528 | 55 | 49

7. Secondary Outcome: Antibody Concentrations for Diphteria Toxoid (D) and Tetanus Toxoid (T)
Description: Anti-D and anti-T antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in International Units per milliliter (IU/mL).
Time Frame: At Day 0 and Month 1 post-Boostrix® vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 713 | 675 | 108 | 104
IU/mL
  Anti-D, Day 0: number analyzed (Participants) | 706 | 670 | 104 | 95
  Anti-D, Day 0 | 0.4 [0.4 to 0.4] | 0.4 [0.3 to 0.4] | 0.2 [0.1 to 0.2] | 0.2 [0.2 to 0.3]
  Anti-D, Month 1: number analyzed (Participants) | 712 | 653 | 106 | 98
  Anti-D, Month 1 | 3.1 [2.8 to 3.5] | 3.4 [3.0 to 3.8] | 1.0 [0.7 to 1.4] | 1.0 [0.6 to 1.4]
  Anti-T, Day 0: number analyzed (Participants) | 711 | 675 | 106 | 104
  Anti-T, Day 0 | 1.5 [1.4 to 1.7] | 1.5 [1.3 to 1.6] | 0.5 [0.4 to 0.7] | 0.6 [0.4 to 0.8]
  Anti-T, Month 1: number analyzed (Participants) | 713 | 654 | 108 | 102
  Anti-T, Month 1 | 6.5 [6.0 to 7.0] | 7.6 [7.0 to 8.2] | 3.4 [2.7 to 4.3] | 3.6 [2.6 to 5.0]

8. Secondary Outcome: Antibody Concentrations for Pertussis Toxoid (PT), Filamentous Hemagglutinin (FHA) and Pertactin (PRN)
Description: as for outcome 3
Time Frame: At Day 0 and Month 1 post-Boostrix® vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 713 | 676 | 108 | 104
EL.U/mL
  Anti-PT, Day 0: number analyzed (Participants) | 703 | 676 | 108 | 104
  Anti-PT, Day 0 | 6.4 [5.9 to 6.9] | 6.5 [6.0 to 7.1] | 8.0 [6.4 to 10.0] | 8.0 [6.4 to 9.9]
  Anti-PT, Month 1: number analyzed (Participants) | 683 | 629 | 103 | 97
  Anti-PT, Month 1 | 57.5 [53.1 to 62.3] | 76.9 [71.1 to 83.2] | 51.2 [40.8 to 64.2] | 59.3 [47.0 to 74.8]
  Anti-FHA, Day 0: number analyzed (Participants) | 705 | 672 | 107 | 103
  Anti-FHA, Day 0 | 36.6 [33.7 to 39.9] | 36.2 [33.2 to 39.5] | 54.5 [43.2 to 68.7] | 59.0 [46.5 to 75.0]
  Anti-FHA, Month 1: number analyzed (Participants) | 712 | 654 | 107 | 100
  Anti-FHA, Month 1 | 467.6 [434.9 to 502.8] | 663.3 [613.3 to 717.4] | 502.5 [409.5 to 616.7] | 669.6 [539.1 to 831.8]
  Anti-PRN, Day 0: number analyzed (Participants) | 713 | 676 | 108 | 103
  Anti-PRN, Day 0 | 12.6 [11.4 to 13.9] | 12.9 [11.7 to 14.3] | 7.5 [5.9 to 9.4] | 6.4 [5.0 to 8.2]
  Anti-PRN, Month 1: number analyzed (Participants) | 713 | 655 | 108 | 101
  Anti-PRN, Month 1 | 234.9 [208.7 to 264.3] | 343.6 [302.5 to 390.1] | 87.9 [60.1 to 128.5] | 97.0 [68.1 to 138.4]

9. Secondary Outcome: Number of Subjects With Booster Response Against Diphteria Toxoid (D) and Tetanus Toxoid (T) Antigens
Description: Booster responses for anti-D and anti-T antibodies are defined as: For initially seronegative subjects [pre-vaccination concentration below (<) cut-off 0.1 IU/mL]: antibody concentrations at least four times the assay cut-off (post-vaccination concentration ≥ 0.4 IU/mL), one month after vaccination with Boostrix®; For initially seropositive subjects (pre-vaccination concentration ≥ 0.1 IU/mL): an increase in antibody concentrations of at least four times the pre-vaccination concentration, one month after vaccination with Boostrix®.
Time Frame: At Month 1 post-Boostrix® vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 710 | 650 | 106 | 102
Participants
  Anti-D: number analyzed (Participants) | 705 | 645 | 103 | 92
  Anti-D | 487 | 459 | 61 | 48
  Anti-T | 293 | 320 | 62 | 63

10. Secondary Outcome: Number of Subjects With Booster Response Against Pertussis Toxoid (PT), Filamentous Hemagglutinin (FHA) and Pertactin (PRN) Antigens
Description: Booster responses for anti-PT, anti-FHA and anti-PRN are defined as: For initially seronegative subjects (pre-vaccination concentration < cut-off of 5 EL.U/mL): antibody concentrations at least four times the cut-off (post-vaccination concentration ≥ 20 EL.U/mL), one month after vaccination with Boostrix®; For initially seropositive subjects with pre-vaccination concentration ≥ 5 EL.U/mL and < 20 EL.U/mL: an increase in antibody concentrations of at least four times the pre-vaccination concentration one month after vaccination with Boostrix®; For initially seropositive subjects with pre-vaccination concentration ≥ 20 EL.U/mL: an increase in antibody concentrations of at least two times the pre-vaccination concentration one month after vaccination with Boostrix®.
Time Frame: At Month 1 post-Boostrix® vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 712 | 652 | 108 | 100
Participants
  Anti-PT: number analyzed (Participants) | 676 | 627 | 103 | 97
  Anti-PT | 514 | 530 | 71 | 68
  Anti-FHA: number analyzed (Participants) | 703 | 647 | 106 | 99
  Anti-FHA | 651 | 621 | 94 | 91
  Anti-PRN | 630 | 589 | 79 | 77

11. Secondary Outcome: Anti-H1N1, Anti-H3N2 and Anti-B Antibody Titers
Description: Anti-H1N1, anti-H3N2 and anti-B antibody titers are presented as geometric mean titers (GMTs).
Time Frame: At Month 1 post-Fluarix® vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 711 | 675 | 108 | 103
Titers
  Anti-H1N1 | 189.1 [171.7 to 208.3] | 181.6 [165.5 to 199.3] | 79.9 [65.0 to 98.3] | 89.3 [72.8 to 109.5]
  Anti-H3N2 | 368.7 [337.9 to 402.3] | 337.3 [309.2 to 367.9] | 333.6 [267.8 to 415.5] | 276.8 [212.4 to 360.8]
  Anti-B | 210.1 [194.4 to 227.0] | 222.8 [205.9 to 241.1] | 221.2 [184.3 to 265.4] | 214.3 [175.4 to 261.8]

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site. Subjects from Boostrix+Fluarix Groups (19-64 YOA and ≥ 65 YOA) received only one vaccination dose (Boostrix® vaccine co-administered with Fluarix® vaccine), at Day 0.
Time Frame: During the 15-day (Day 0-14) period following each dose and across doses, up to 2 months
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and with the symptom sheet filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 725 | 710 | 110 | 108
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 725 | 707 | 110 | 108
  Any Pain, Dose 1 | 467 | 315 | 41 | 25
  Grade 3 Pain, Dose 1: number analyzed (Participants) | 725 | 707 | 110 | 108
  Grade 3 Pain, Dose 1 | 28 | 7 | 0 | 1
  Any Redness, Dose 1: number analyzed (Participants) | 725 | 707 | 110 | 108
  Any Redness, Dose 1 | 180 | 148 | 23 | 15
  Grade 3 Redness, Dose 1: number analyzed (Participants) | 725 | 707 | 110 | 108
  Grade 3 Redness, Dose 1 | 4 | 5 | 3 | 2
  Any Swelling, Dose 1: number analyzed (Participants) | 725 | 707 | 110 | 108
  Any Swelling, Dose 1 | 179 | 93 | 18 | 11
  Grade 3 Swelling, Dose 1: number analyzed (Participants) | 725 | 707 | 110 | 108
  Grade 3 Swelling, Dose 1 | 12 | 7 | 3 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 0 | 664 | 0 | 104
  Any Pain, Dose 2 | 0 | 327 | 0 | 30
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 0 | 664 | 0 | 104
  Grade 3 Pain, Dose 2 | 0 | 9 | 0 | 3
  Any Redness, Dose 2: number analyzed (Participants) | 0 | 664 | 0 | 104
  Any Redness, Dose 2 | 0 | 124 | 0 | 16
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 0 | 664 | 0 | 104
  Grade 3 Redness, Dose 2 | 0 | 3 | 0 | 2
  Any Swelling, Dose 2: number analyzed (Participants) | 0 | 664 | 0 | 104
  Any Swelling, Dose 2 | 0 | 106 | 0 | 9
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 0 | 664 | 0 | 104
  Grade 3 Swelling, Dose 2 | 0 | 6 | 0 | 0
  Any Pain, Across doses | 467 | 429 | 41 | 44
  Grade 3 Pain, Across doses | 28 | 15 | 0 | 4
  Any Redness, Across doses | 180 | 207 | 23 | 20
  Grade 3 Redness, Across doses | 4 | 8 | 3 | 4
  Any Swelling, Across doses | 179 | 160 | 18 | 17
  Grade 3 Swelling, Across doses | 12 | 12 | 3 | 1

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal (nausea, vomiting, diarrhoea and/or abdominal pain), headache, joint pain, muscle aches and shivering. Any = occurrence of the symptom regardless of intensity grade or relationship to the study vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination. Subjects from Boostrix+Fluarix Groups (19-64 YOA and ≥ 65 YOA) received only one vaccination dose (Boostrix® vaccine co-administered with Fluarix® vaccine), at Day 0.
Time Frame: During the 15-day (Day 0-14) period following each dose and across doses, up to 2 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 726 | 710 | 110 | 108
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Any Fatigue, Dose 1 | 220 | 165 | 20 | 18
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Grade 3 Fatigue, Dose 1 | 22 | 15 | 0 | 1
  Related Fatigue, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Related Fatigue, Dose 1 | 144 | 103 | 15 | 12
  Any Fever, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Any Fever, Dose 1 | 54 | 52 | 4 | 3
  Grade 3 Fever, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Grade 3 Fever, Dose 1 | 1 | 0 | 0 | 0
  Related Fever, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Related Fever, Dose 1 | 28 | 28 | 3 | 2
  Any Gastrointestinal, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Any Gastrointestinal, Dose 1 | 121 | 101 | 18 | 12
  Grade 3 Gastrointestinal, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Grade 3 Gastrointestinal, Dose 1 | 16 | 11 | 2 | 1
  Related Gastrointestinal, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Related Gastrointestinal, Dose 1 | 68 | 55 | 12 | 6
  Any Headache, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Any Headache, Dose 1 | 225 | 197 | 17 | 17
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Grade 3 Headache, Dose 1 | 24 | 25 | 2 | 1
  Related Headache, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Related Headache, Dose 1 | 143 | 118 | 12 | 13
  Any Joint pain, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Any Joint pain, Dose 1 | 137 | 87 | 14 | 13
  Grade 3 Joint pain, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Grade 3 Joint pain, Dose 1 | 10 | 10 | 0 | 0
  Related Joint pain, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Related Joint pain, Dose 1 | 97 | 56 | 8 | 12
  Any Muscle aches, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Any Muscle aches, Dose 1 | 266 | 193 | 26 | 18
  Grade 3 Muscle aches, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Grade 3 Muscle aches, Dose 1 | 27 | 15 | 2 | 0
  Related Muscle aches, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Related Muscle aches, Dose 1 | 194 | 131 | 16 | 17
  Any Shivering, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Any Shivering, Dose 1 | 70 | 44 | 5 | 4
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Grade 3 Shivering, Dose 1 | 8 | 5 | 0 | 0
  Related Shivering, Dose 1: number analyzed (Participants) | 726 | 707 | 110 | 108
  Related Shivering, Dose 1 | 42 | 30 | 4 | 3
  Any Fatigue, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Any Fatigue, Dose 2 | 0 | 115 | 0 | 6
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Grade 3 Fatigue, Dose 2 | 0 | 18 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Related Fatigue, Dose 2 | 0 | 83 | 0 | 5
  Any Fever, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Any Fever, Dose 2 | 0 | 38 | 0 | 4
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Grade 3 Fever, Dose 2 | 0 | 1 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Related Fever, Dose 2 | 0 | 23 | 0 | 2
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Any Gastrointestinal, Dose 2 | 0 | 55 | 0 | 3
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Grade 3 Gastrointestinal, Dose 2 | 0 | 6 | 0 | 1
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Related Gastrointestinal, Dose 2 | 0 | 29 | 0 | 1
  Any Headache, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Any Headache, Dose 2 | 0 | 132 | 0 | 8
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Grade 3 Headache, Dose 2 | 0 | 12 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Related Headache, Dose 2 | 0 | 87 | 0 | 7
  Any Joint pain, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Any Joint pain, Dose 2 | 0 | 75 | 0 | 7
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Grade 3 Joint pain, Dose 2 | 0 | 14 | 0 | 0
  Related Joint pain, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Related Joint pain, Dose 2 | 0 | 52 | 0 | 7
  Any Muscle aches, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Any Muscle aches, Dose 2 | 0 | 183 | 0 | 14
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Grade 3 Muscle aches, Dose 2 | 0 | 21 | 0 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Related Muscle aches, Dose 2 | 0 | 150 | 0 | 13
  Any Shivering, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Any Shivering, Dose 2 | 0 | 48 | 0 | 2
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Grade 3 Shivering, Dose 2 | 0 | 7 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 0 | 665 | 0 | 104
  Related Shivering, Dose 2 | 0 | 34 | 0 | 2
  Any Fatigue, Across doses | 220 | 218 | 20 | 22
  Grade 3 Fatigue, Across doses | 22 | 30 | 0 | 1
  Related Fatigue, Across doses | 144 | 149 | 15 | 16
  Any Fever, Across doses | 54 | 80 | 4 | 7
  Grade 3 Fever, Across doses | 1 | 1 | 0 | 0
  Related Fever, Across doses | 28 | 47 | 3 | 4
  Any Gastrointestinal, Across doses | 121 | 132 | 18 | 13
  Grade 3 Gastrointestinal, Across doses | 16 | 16 | 2 | 2
  Related Gastrointestinal, Across doses | 68 | 73 | 12 | 7
  Any Headache, Across doses | 225 | 251 | 17 | 22
  Grade 3 Headache, Across doses | 24 | 33 | 2 | 1
  Related Headache, Across doses | 143 | 163 | 12 | 19
  Any Joint pain, Across doses | 137 | 135 | 14 | 18
  Grade 3 Joint pain, Across doses | 10 | 23 | 0 | 0
  Related Joint pain, Across doses | 97 | 89 | 8 | 17
  Any Muscle aches, Across doses | 266 | 287 | 26 | 26
  Grade 3 Muscle aches, Across doses | 27 | 34 | 2 | 0
  Related Muscle aches, Across doses | 194 | 224 | 16 | 25
  Any Shivering, Across doses | 70 | 80 | 5 | 5
  Grade 3 Shivering, Across doses | 8 | 10 | 0 | 0
  Related Shivering, Across doses | 42 | 56 | 4 | 4

14. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day period (Day 0-30) following each vaccination, up to 2 months
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 748 | 749 | 112 | 109
Participants | 161 | 205 | 22 | 21

15. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Throughout the whole study period (from Day 0 to Month 2)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix+Fluarix 19-64 YOA Group | Fluarix Boostrix 19-64 YOA Group | Boostrix+Fluarix ≥ 65 YOA Group | Fluarix Boostrix ≥ 65 YOA Group
Number analyzed (Participants) | 748 | 749 | 112 | 109
Participants | 2 | 7 | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 15-day (Day 0-14) period following each vaccination; Unsolicited AEs: during the 31-day period (Day 0-30) following each vaccination; SAEs: throughout the whole study period (from Day 0 to Month 2).
Arm/Group | Boostrix+Fluarix Group | Fluarix Boostrix Group
All-Cause Mortality (participants affected / at risk) | 0/860 | 0/858
Serious Adverse Events (participants affected / at risk) | 3/860 | 7/858
Other Adverse Events (participants affected / at risk) | 640/860 | 619/858
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix+Fluarix Group (N=860) | Fluarix Boostrix Group (N=858)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix+Fluarix Group (N=860) | Fluarix Boostrix Group (N=858)
Arthralgia (Musculoskeletal and connective tissue disorders) | 151 (152) | 156 (186)
Chills (General disorders) | 76 (76) | 86 (99)
Erythema (Skin and subcutaneous tissue disorders) | 203 (203) | 227 (303)
Fatigue (General disorders) | 240 (240) | 240 (306)
Gastrointestinal disorder (Gastrointestinal disorders) | 139 (139) | 145 (171)
Headache (Nervous system disorders) | 244 (244) | 276 (361)
Myalgia (Musculoskeletal and connective tissue disorders) | 294 (294) | 313 (411)
Pain (General disorders) | 509 (513) | 473 (698)
Pyrexia (General disorders) | 59 (59) | 88 (98)
Swelling (General disorders) | 198 (198) | 177 (219)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.